CLINICAL TRIAL: NCT02786264
Title: Pilot Analysis of the Association Between Types of Anesthetic and Outcomes in Transfemoral Aortic Valve Replacement
Brief Title: Association of Type of Anesthetic and Outcomes in Transfemoral Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1604017590
Record Dates: First submitted 2016-05-11; First posted 2016-05-30 (Estimated); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2022-08

CONDITIONS: Aortic Stenosis
Keywords: transcatheter aortic valve replacement; anesthesia; conscious sedation; managed anesthesia care
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Propofol-dominant Sedation: Patients receiving propofol infusion for TAVR as the primary drug for sedation.
  Interventions: Drug: Propofol
- Dexmedetomidine-dominant Sedation: Patients receiving dexmedetomidine infusion for TAVR as the primary drug for sedation.
  Interventions: Drug: Dexmedetomidine with propofol; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine with propofol — A dexmedetomidine- dominant anesthetic will be defined as an anesthetic that included a continuous infusion of dexmedetomidine within 15 minutes of anesthesia start. This group was subsequently modified in light of retrospective data collection to specify a group receiving dexmedetomidine in combination with propofol.
  Other Names: Precedex
  Groups: Dexmedetomidine-dominant Sedation
Drug: Propofol — A propofol-dominant anesthetic will be defined as an anesthetic that included a continuous infusion of propofol within 15 minutes of anesthesia start. This definition was subsequently modified to include patients who received propofol infusion but not dexmedetomidine.
  Other Names: Diprivan

SUMMARY:
This study proposes to perform a descriptive analysis and pilot observational study looking at the types and quantity of anesthetic agents used and their associations with outcomes among patients scheduled to receive transfemoral aortic valve replacements (TAVR) at Yale New Haven Hospital (YNHH).

DETAILED DESCRIPTION:
This study proposes to perform a descriptive analysis and pilot observational study looking at the types and quantity of anesthetic agents used and their associations with outcomes among patients scheduled to receive TAVR at YNHH.

Hypothesis 1: TAVR surgery done under monitored anesthesia care are performed using some combination of the following anesthetics: dexmedetomidine, propofol, fentanyl, and midazolam.

Hypothesis 2: Age-adjusted dosing of these agents will be insufficient to account for extreme age after controlling for preoperative comorbid status.

Hypothesis 3: The rate of conversion to general anesthesia will be unrelated to the type of conscious sedation used.

Hypothesis 4: ICU length of stay, delirium, hospital length of stay, and length of hospital stay will be shorter for patients who were sedated using dexmedetomidine vs those without.

Research Plan: The research will be done via chart review and analysis of data already contained in the Multicenter Perioperative Outcomes Group databases at Yale. The possible risks are primarily the risk to privacy that is inherent in any retrospective chart review. The benefit may be to suggest areas of future study to improve sedation practices for TAVR at Yale and elsewhere. Information recorded will include demographic and preoperative medical assessment from prior to the TAVR, the anesthetic record, and the post-operative course of recovery for patients undergoing TAVR. These data will include age, gender, comorbidities, laboratory values, vital signs, and the results of imaging studies as well as other records potentially related to the above hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent TAVR at YNHH under planned conscious sedation with monitored anesthetic care

Exclusion Criteria:

* Patients who received monitored anesthesia care without the receipt of any study intervention drug (propofol, fentanyl, midazolam, or dexmedetomidine).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent TAVR under a plan for conscious sedation with monitored anesthetic care rather than general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schonberger, MD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frohlich GM, Lansky AJ, Webb J, Roffi M, Toggweiler S, Reinthaler M, Wang D, Hutchinson N, Wendler O, Hildick-Smith D, Meier P. Local versus general anesthesia for transcatheter aortic valve implantation (TAVR)--systematic review and meta-analysis. BMC Med. 2014 Mar 10;12:41. doi: 10.1186/1741-7015-12-41. PMID 24612945
- Available data/document: Statistical Analysis Plan — https://docs.google.com/document/d/1SUzYG_9aKT5sSkPXEmhvRTqvhXRflQLBiXJe59inDh4/edit?usp=sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a retrospective chart review and did not include prospective enrollment. As noted in the pre-assignment details, the number of enrolled participants was determined by chart review.
Pre-assignment Details: As specified above, this study was a retrospective chart review and thus enrollment was determined by existence of charts rather than by prospective enrollment. While patients were screened for other modes of sedation, data were only collected on the two groups included presently.
Groups:
- Propofol-dominant Sedation: Patients receiving propofol infusion for TAVR as the primary drug for sedation.
  Propofol: A propofol-dominant anesthetic will be defined as an anesthetic that included a continuous infusion of propofol within 15 minutes of anesthesia start.
- Propofol With Dexmedetomidine Group: Patients who qualified for Both the Propofol Dominant and the Dexmedetomidine Dominant group were categorized into this fourth group.
Period: Overall Study
Arm/Group | Propofol-dominant Sedation | Propofol With Dexmedetomidine Group
Started | 39 | 34
Completed | 39 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was not a clinical trial but rather a retrospective observational study in which arms were developed based on an understanding of the descriptive data. As stated in the manuscript, "As the dexmedetomidine-dominant and fentanyl-dominant groups had limited sample size, the authors decided to focus on the propofol-dominant and dexmedetomidine plus propofol groups for analysis of outcomes."
Groups:
- Propofol and Dexmedetomidine: Defined as any MAC that included both propofol and dexmedetomidine and may have included fentanyl, remifentanil, or midazolam
- Propofol Only: Defined as any MAC that included propofol infusions or injections in the absence of dexmedetomidine. These patients also may have received injections of fentanyl, remifentanil, or midazolam.
- Total: Total of all reporting groups
Arm/Group | Propofol and Dexmedetomidine | Propofol Only | Total
Number analyzed (Participants) | 34 | 39 | 73
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 84 [78 to 88] | 87 [81 to 90] | 87 [80 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 14 | 24 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 31 | 34 | 65
  Black | 1 | 1 | 2
  Hispanic/Latino | 1 | 2 | 3
  Other | 1 | 0 | 1
  Unknown | 0 | 2 | 2
Height [Median (Inter-Quartile Range); unit: meters] | 1.6 [1.6 to 1.7] | 1.6 [1.6 to 1.7] | 1.6 [1.6 to 1.7]
Weight [Median (Inter-Quartile Range); unit: kg] | 71.5 [59.1 to 80.5] | 76.6 [65.6 to 85.1] | 73.7 [62 to 83.2]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 25.6 [22.1 to 29.3] | 29.2 [23.9 to 32.3] | 26.7 [23.9 to 30.7]
American Society of Anesthesiologists (ASA) Physical Status Score [Count of Participants; unit: Participants] — ASA Physical Status is a measure of comorbidity developed by the American Society of Anesthesiologists. It is graded ordinally from 1 to 6 whereby 1 represents a healthy patient, 4 a patient with serious systemic disease, 5 a moribund patient, and 6 a brain dead individual presenting for organ donation after death.
  Participants
    3 | 5 | 3 | 8
    4 | 29 | 36 | 65
New York Heart Association Congestive Heart Failure (NYHA CHF)HF classification [Count of Participants; unit: Participants] — NYHA CHF is graded from 1 to 4 in which 1 is a person without heart failure, 2 is a person with sympoms only during exercise, and 3 iand 4 are progressively more serious stages of heart failure.
  Participants
    2 | 5 | 1 | 6
    3 | 24 | 32 | 56
    4 | 5 | 6 | 11
Left ventricular ejection fraction (LVEF) [Median (Inter-Quartile Range); unit: %] | 63 [59 to 67] | 62 [55 to 66] | 62 [55 to 66]
Alcoholism [Count of Participants; unit: Participants]
  No | 34 | 38 | 72
  Yes | 0 | 1 | 1
Anxiety disorder [Count of Participants; unit: Participants]
  No | 30 | 35 | 65
  Yes | 4 | 4 | 8
Atrial fibrillation [Count of Participants; unit: Participants]
  No | 22 | 18 | 40
  Yes | 12 | 21 | 33
Cerebrovascular disease [Count of Participants; unit: Participants]
  No | 29 | 38 | 67
  Yes | 5 | 1 | 6
Congestive Heart Failure (CHF) [Count of Participants; unit: Participants]
  No | 15 | 17 | 32
  Yes | 19 | 22 | 41
Coronary Artery Disease (CAD) [Count of Participants; unit: Participants]
  No | 12 | 13 | 25
  Yes | 22 | 26 | 48
Diabetes [Count of Participants; unit: Participants]
  No | 24 | 27 | 51
  Yes | 10 | 12 | 22
Hypertension [Count of Participants; unit: Participants]
  No | 4 | 5 | 9
  Yes | 30 | 34 | 64
Depression [Count of Participants; unit: Participants]
  No | 30 | 35 | 65
  Yes | 4 | 4 | 8
Obstructive sleep apnea [Count of Participants; unit: Participants]
  No | 32 | 33 | 65
  Yes | 2 | 6 | 8
Peripheral vascular disease [Count of Participants; unit: Participants]
  No | 27 | 35 | 62
  Yes | 7 | 4 | 11
Psychosis [Count of Participants; unit: Participants]
  No | 34 | 39 | 73
  Yes | 0 | 0 | 0
Renal disease [Count of Participants; unit: Participants]
  No | 22 | 30 | 52
  Yes | 12 | 9 | 21
Substance abuse [Count of Participants; unit: Participants]
  No | 34 | 39 | 73
  Yes | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Procedure Length
Description: Procedure length will be collected from retrospective analysis of charts.
Time Frame: During surgery
Population: NB: The analyzed groups are the subset of the participant arms that were deemed to have sufficient numbers for comparison. Other groups were excluded from analysis after descriptive understanding of the makeup of this retrospective cohort.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Propofol and Dexmedetomidine | Propofol Only
Number analyzed (Participants) | 34 | 39
minutes | 114.5 [102 to 137] | 100 [87 to 123]

2. Secondary Outcome: ICU Length of Stay
Description: ICU length of stay will be collected from retrospective analysis of charts.
Time Frame: From the conclusion of surgery until patient leaves the ICU, up to 2 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Propofol and Dexmedetomidine | Propofol Only
Number analyzed (Participants) | 34 | 39
days | 1 [1 to 1] | 1 [1 to 2]

3. Secondary Outcome: Rate of Conversion to General Anesthesia
Description: Rate of conversion to general anesthesia will be collected from retrospective analysis of charts.
Time Frame: During surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol and Dexmedetomidine | Propofol Only
Number analyzed (Participants) | 34 | 39
Participants
  No | 31 | 38
  Yes | 3 | 1

4. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay will be collected via retrospective analysis of charts.
Time Frame: From the conclusion of surgery until patient is discharged, up to 2 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Propofol and Dexmedetomidine | Propofol Only
Number analyzed (Participants) | 34 | 39
days | 2 [2 to 3] | 2 [2 to 3]

5. Secondary Outcome: Delirium Incidence
Description: Whether or not the patient experiences delirium during their hospital stay as recorded in their notes by the treating physician.
Time Frame: From the conclusion of surgery until patient is discharged, up to 2 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol and Dexmedetomidine | Propofol Only
Number analyzed (Participants) | 34 | 39
Participants
  No | 34 | 38
  Yes | 0 | 1

ADVERSE EVENTS:
Time Frame: Retrospective study. No adverse events.
Description: Retrospective study. No adverse events.
Groups:
- Propofol and Dexmedetomidine: Defined as any MAC that included both propofol and dexmedetomidine and may have included fentanyl, remifentanil, or midazolam.
  NB: The analyzed groups are the subset of the participant arms that were deemed to have sufficient numbers for comparison. Other groups were excluded from analysis after descriptive understanding of the makeup of this retrospective cohort.
- Propofol Only: Defined as any MAC that included propofol infusions or injections in the absence of dexmedetomidine. These patients also may have received injections of fentanyl, remifentanil, or midazolam.
  NB: The analyzed groups are the subset of the participant arms that were deemed to have sufficient numbers for comparison. Other groups were excluded from analysis after descriptive understanding of the makeup of this retrospective cohort.
Arm/Group | Propofol and Dexmedetomidine | Propofol Only
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02786264/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT02786264/SAP_001.pdf